CLINICAL TRIAL: NCT02330445
Title: Phase I/II Open Label Evaluation of Safety and Feasibility of 6 Months IV PRTX-100 Administrations in Previous Rheumatoid Arthritis Study Participants and Development of Immunological Samples for Assay Development From Normal Volunteers
Brief Title: 6-Month Phase I/II Open Label PRTX-100 in Previous Rheumatoid Arthritis Study Participants and Sera Collection
Acronym: SPARTA-II
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Protalex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRTX-100-105
Record Dates: First submitted 2014-12-18; First posted 2015-01-05 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Staphylococcal Protein A

STUDY DESIGN:
Intervention Model Description: Two parts of recipients are assigned for this Phase I/II open label, single site study. Part A subjects are all who had RA while Part B subjects are healthy volunteers. All subject are allocated to the single treatment group at a fixed dose of 6.0μg/kg of IV PRTX-100.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Experimental): Up to 12 Part A recipients will have rheumatoid arthritis since this was an entry criterion for Study 104. All subjects will be allocated to the single treatment group at a fixed dose of 6 μg/kg of IV PRTX-100. Subjects will receive four weekly doses followed by 5 monthly doses of PRTX-100. Since subjects will be followed for 28 days after their last dose, the total duration of the study is approximately 8 months. Subjects will be evaluated for adverse events, rheumatoid arthritis activity and the development of anti-PRTX-100 antibodies. The feasibility of different assessment methods of disease activity may be explored. Novel methods of joint evaluation will be explored. Adverse events will be evaluated for at least four weeks after the last dose of PRTX-100.
  Interventions: Drug: PRTX-100
- Part B (Experimental): Five healthy subjects will be allocated to the single treatment group at a fixed dose of 6 μg/kg of IV PRTX-100. Subjects will receive four weekly doses. All subjects will have a serum collection requiring approximately 600 mL of blood. Since subjects will be followed for 28 days after their last dose, the total duration of the study is approximately 3 months. Subjects will be evaluated for adverse events and the development of anti-PRTX-100 antibodies. Adverse events will be evaluated for at least four weeks after the last dose of PRTX-100.
  Interventions: Drug: PRTX-100

INTERVENTIONS:
Drug: PRTX-100 — 6 micrograms PRTX-100 per kilogram of body weight administered via infusion
  Other Names: SpA; Staphylococcal Protein A

SUMMARY:
Part A Primary Objective To determine the safety of six months of PRTX-100 administration. Part B Primary Objective To obtain antisera from normal volunteers that have developed anti-PRTX-100 antibodies.

Secondary Objective(s) To assess rheumatoid arthritis activity during the period of PRTX-100 treatment To evaluate the development of anti-PRTX-100 antibodies To explore feasibility of joint evaluations with ultrasound To explore feasibility of biomarkers as disease markers

DETAILED DESCRIPTION:
Although the majority of RA patients achieve an amelioration of their RA with older disease modifying agents such as methotrexate and leflunomide, all of these agents provoke adverse events. The newer more active biological agents have a distinct safety profile that includes an increased risk of serious infections. They have an annual treatment expense in the tens of thousands of dollars a year. PRTX-100 may be able to modify the disease course of rheumatoid arthritis with an improved safety profile compared to available agents and a dosing regimen comparable to the therapies currently available. This study is done to describe the adverse event profile of 6 μg/kg of PRTX-100 administered IV for longer periods of treatment that might be required for RA therapy. Secondary objectives include: evaluation of the clinical response of subjects with previous administration of PRTX-100; evaluation of anti-PRTX antibody presence and effect on activity; evaluation of "Power Doppler" ultrasound in the assessment of joint inflammation; and evaluation of biomarkers.

Assay development is an intrinsic part of drug and biological development. The current assay for anti-PRTX-100 antibodies depends on a very limited supply of serum available from individuals in early trials. It will be necessary to obtain adequate antisera to provide immunological reagents for this assay. It is not known whether the character of anti-PRTX-100 antibodies from volunteers is similar to those produced by patients with immunological disorders on cytotoxic therapy. Antisera will be developed in normal volunteers. The anti-PRTX-100 antibody assay will need to be standardized with a new anti-PRTX-100 antibody source compared to the present human reagent.

ELIGIBILITY:
Part A Inclusion Criteria:

1. Has completed the written informed consent process
2. Received PRTX-100 or placebo in Study 104
3. Receiving methotrexate or leflunomide therapy for at least 12 weeks
4. Must be on a stable weekly dose of methotrexate (12.5 to 25 mg) or daily leflunomide (10-20 mg/day) by the same route of administration for at least 3 weeks prior to the start of study drug.
5. Agrees to notify the investigator when deviating from protocol requirements for concomitant medications
6. Agrees to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study
7. Agrees to avoid elective surgery for the full duration of the study
8. For female subjects: agrees to avoid pregnancy from 28 days prior to Study Day 0 and for the full duration of the study. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD), or the combination of a condom or diaphragm with spermicide.

Part A Exclusion Criteria:

1. Diagnosis of any other inflammatory arthritis (e.g. psoriatic arthritis, spondyloarthropathy, gout)
2. ACR Functional Classification IV
3. Systemic involvement secondary to rheumatoid arthritis (vasculitis, pulmonary fibrosis or Felty's syndrome. Secondary Sjogren's syndrome is permitted.
4. Any receipt of abatacept, adalimumab, certolizumab pegol, etanercept, golimumab, tocilizumab or tofacitinib within 3 weeks of Study Day 0
5. Any receipt of infliximab within 6 weeks of Study Day 0
6. Any receipt of rituximab or other anti-CD20 antibodies within 12 months of study day 0
7. Any receipt of another investigational product within 4 weeks or 4 half-lives whichever is longer prior to Study Day 0
8. Hepatitis B surface antigen positive, HIV positive, hepatitis C antibody positive
9. Uncontrolled Type 2 Diabetes or Type I diabetes
10. Positive urine pregnancy test
11. Diagnosis of hepatic cirrhosis
12. Urinalysis must reflect no evidence of systemic or local disease process
13. Severe anemia, defined as < 10 g/dL or hematocrit < 30%
14. Evidence of significant active infection
15. Shared a residence within the last year with an individual on anti-tuberculosis treatment or with culture or smear positive tuberculosis
16. Previous medical history that may compromise the safety of the subject in the study, including but not limited to: severe impairment of pulmonary function or other pulmonary disease; chronic illness with signs of cardiac or renal failure; suspected progressive neurological disease or poorly controlled epilepsy
17. Evidence of a new acute illness that may compromise the safety of the subject in the study
18. History or evidence on physical examination of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the safety of the study drug
19. History or evidence (including chest X-ray) of active tuberculosis
20. Any current medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the subject will comply with the protocol.

Part B Inclusion Criteria

1. Has completed the written informed consent process
2. Is in a state of good health
3. Agrees to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study
4. Agrees to avoid elective surgery for the full duration of the study
5. For female subjects: agrees to avoid pregnancy from 28 days prior to Study Day 0 and for the full duration of the study. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD), or the combination of a condom or diaphragm with spermicide.

Part B Exclusion Criteria

1. Diagnosis of cancer or autoimmune disease.
2. Any receipt of another investigational product within 4 weeks or 4 half-lives whichever is longer prior to Study Day 0
3. Hepatitis B surface antigen positive, HIV positive, hepatitis C antibody positive
4. Uncontrolled Type 2 Diabetes or Type I diabetes
5. Diagnosis of hepatic cirrhosis
6. Positive urine pregnancy test
7. Urinalysis must reflect no evidence of systemic or local disease process
8. Severe anemia, defined as < 10 g/dL or hematocrit < 30%
9. Previous medical history that may compromise the safety of the subject in the study, including but not limited to: severe impairment of pulmonary function or other pulmonary disease; chronic illness with signs of cardiac or renal failure; suspected progressive neurological disease or poorly controlled epilepsy
10. Evidence of a new acute illness that may compromise the safety of the subject in the study
11. History or evidence on physical examination of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the safety of the study drug
12. Any current medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the subject will comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04-18 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Safety (Analysis of Adverse Events) | 6 months
  Number, severity, and attribution of relatedness of Adverse Events will be analyzed.

SECONDARY OUTCOMES:
ACR-28 joint count | 6 months
  ACR 28-joint counts (number of tender and swollen joints) will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
Patient's global assessment of disease activity | 6 months
  Patient's global assessment of disease activity (0-10) will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
Patient's assessment of pain VAS | 6 months
  Patient's assessment of pain VAS (0-10) will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
Physician's global assessment of disease activity | 6 months
  Physician's global assessment of disease activity (0-10) will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
MDHAQ - Physical Function | 6 months
  MDHAQ Physical Function (0-10) will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
MDHAQ - Joint Pain | 6 months
  MDHAQ Joint Pain (0-48) will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
MDHAQ - Fatigue | 6 months
  MDHAQ Fatigue (0-10) will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
RAPID 3 | 6 months
  RAPID 3 (0-30) will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
CDAI | 6 months
  Clinical Disease Activity Index (0-76) will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
DAS28-CRP | 6 months
  DAS28-CRP (0-10) will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
hsCRP | 6 months
  C-Reactive Protein (hsCRP) lab values (mg/dL) will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
ESR | 6 months
  Erythrocyte Sedimentation Rate (mm/hr) will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
Biomarker Correlation | 6 months
  Vectra-DA scores (1-100) will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
Disease activity | 6 months
  ACR 28-joint counts (tender and swollen), patient's global assessment of disease activity, patient's assessment of pain VAS, physician's global assessment of disease activity, MDHAQ (overall, physical function, joint pain, and fatigue), RAPID 3, CDAI, DAS28-CRP, CRP, ESR, Vectra-DA, and UPD joint counts, will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
Ultrasound Power Doppler Joint Count | 6 months
  UPD joint counts (0-36) will be summarized descriptively by assessment time point in addition to change and percent change from baseline values, as well as in categorical analyses for disease activity.
Immunogenicity | 6 months
  The occurrence of anti-PRTX-100 antibodies (positive/negative) will be summarized descriptively for the observed values and change from baseline results.

OTHER OUTCOMES:
Sera Collection | 77 Days
  To obtain antisera from normal volunteers that have developed anti-PRTX-100 antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: John B McClain, MD, Study Director — Protalex, Inc.
Locations (1):
- Protalex Investigational Site, Coeur d'Alene, Idaho, United States

IPD SHARING:
Plan to Share IPD: No